CLINICAL TRIAL: NCT02768792
Title: LCCC 1522: Phase 2 Study of High Dose Cytarabine Followed by Pembrolizumab in Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: High Dose Cytarabine Followed by Pembrolizumab in Relapsed/Refractory AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1522
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label, multicenter, single-arm (Other): Pembrolizumab 200 mg is administered IV once as monotherapy, 14 days after the initiation of HiDAC salvage induction chemotherapy. Patients who have a response (i.e., PR/CR/CRi) to induction phase will receive maintenance pembrolizumab at 200 mg IV every 3 weeks for up to 2-years of maintenance therapy (i.e., beginning on day 1 of maintenance). Patients who are ineligible for pembrolizumab administration by day 21 will be removed from the study.
  Interventions: Drug: pembrolizumab,

INTERVENTIONS:
Drug: pembrolizumab, — Pembrolizumab 200 mg is administered IV once as monotherapy, 14 days after the initiation of HiDAC salvage induction chemotherapy. Patients who have a response (i.e., PR/CR/CRi) to induction phase will receive maintenance pembrolizumab at 200 mg IV every 3 weeks for up to 2 years of maintenance therapy (i.e., beginning on day 1 of maintenance).
  Other Names: KEYTRUDA; MK-3475

SUMMARY:
Rationale:The purpose of this research study is to test the effectiveness of the standard high dose cytarabine (HiDAC) on days 1 through 5 followed by a single dose of pembrolizumab on day 14 as induction therapy in patients with relapsed and refractory acute myeloid leukemia (AML). Patients who achieve a response to treatment will continue on the study drug (pembrolizumab) every 3 weeks for up to 2 years maintenance therapy.

Purpose:This is a study about a new investigative drug, pembrolizumab (MK-3475) that is being studied in a clinical research trial together with standard chemotherapy (HiDAC) in relapsed and refractory AML. The study will also explore the association between potential immune biomarkers and clinical outcomes with pembrolizumab; therefore all patients will have blood and bone marrow samples collected before and after treatment to determine the dynamic nature of immune signatures pre and post-treatment.

DETAILED DESCRIPTION:
Primary Objective

1. Estimate the objective overall rate of CR (CR+CRi) for age-adjusted HiDAC (age <60 years: 2 gm/m2 IV Q12hours days 1-5; age >60 years: 1.5 gm/m2 IV Q12hours days 1-5) followed by pembrolizumab 200 mg IV on day 14 in relapsed and refractory AML patients

Secondary Objectives

1. Estimate the rate of unacceptable toxicity associated with HiDAC followed by pembrolizumab as induction therapy
2. Estimate the objective overall response rates (PR+CR+CRi) for HiDAC followed by pembrolizumab.
3. Characterize the toxicity associated with HiDAC followed by pembrolizumab as induction therapy
4. Characterize the toxicity associated with pembrolizumab 200 mg IV Q3weeks when used as monotherapy maintenance after an initial response to induction phase HiDAC followed by pembrolizumab
5. Estimate the relapse-free survival (RFS) and progression-free survival (PFS) of patients receiving maintenance pembrolizumab
6. Estimate the overall survival (OS) of patients who received induction phase treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent for the trial
2. > 18 years and < 70 years of age on day of signing informed consent
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
4. Have histologically or cytologically confirmed recurrent AML as defined by ≥5 % myeloblasts in the bone marrow aspirate and or biopsy.
5. Must have received at least 1 cycle of induction therapy for front-line AML including cytarabine continuous infusion + anthracycline +/- cladribine or etoposide for 1 or 2 cycles, or liposomal cytarabine and daunorubicin (CPX-351), or high dose cytarabine with or without fludarabine, cladribine or clofarabine, > 4 cycles of azacitidine/decitabine or the equivalent experimental therapy (the latter as confirmed by the PI)
6. Cytoreduction allowed with hydroxyurea and/or leukapheresis for up to 14 days prior to D1 of treatment under LCCC1522. Patients must be off hydroxyurea for > 12 hours prior to D1 of treatment under LCCC1522
7. Demonstrate adequate organ function as defined below. All screening labs should be performed within 14 days of D1 of treatment under LCCC1522.

   Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl)-- ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN unless due to Gilbert's Disease, hemolysis or leukemic infiltration OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN Aspartate Aminotransferase (AST)(SGOT) and Alanine Aminotransferase (ALT) (SGPT) ≤ 5 X ULN International Normalized Ratio (INR) or Prothrombin Time (PT)- ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants or patient has disseminated intravascular coagulation deemed by investigator to be due to leukemia Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants or patient has disseminated intravascular coagulation deemed by investigator to be due to leukemia
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of HiDAC treatment and again prior to D1 of pembrolizumab treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. The two birth control methods can be two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from the screening visit throughout the study period up to 120 days after the last dose of study therapy.

   Note: Abstinence is acceptable if this is the usual lifestyle preferred contraception for the subject.
10. Male subjects must agree to use an adequate method of contraception starting with D1 of HiDAC through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of HiDAC treatment. Note: use of steroid eye drops starting at the time of HiDAC administration is allowed.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to pembrolizumab or any of its excipients
5. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has known active central nervous system (CNS) leukemia; subjects with previously treated CNS disease may participate provided they are stable (without evidence of active disease by imaging for at least 4 weeks prior to the first dose of treatment, and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to D1 of treatment.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has evidence of interstitial lung disease or a history of ( non-infectious) pneumonitis that required steroids or current pneumonitis.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
15. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
16. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA qualitative is detected).
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed
18. Has uncontrolled intercurrent illness including, but not limited to, active and uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, and uncontrolled symptomatic cardiac arrhythmia. Patients with infection under active treatment and controlled with antibiotics are eligible.
19. Diagnosed with acute promyelocytic leukemia (APL, M3)
20. Receipt of previous allogeneic stem cell transplant; receipt of previous autologous transplant for AML or non-AML condition is allowed

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Zeidner, MD, Principal Investigator — Lineberger Comprehensive Cancer Center University of North Carolina
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: Web address for UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two cancer centers between August 2016 and April 2019.
Pre-assignment Details: A total of 62 subjects were consented to screen for eligibility. Of these, 19 were determined to be ineligible and 5 withdrew consent prior to starting the study.
Groups:
- Single Arm Pembrolizumab: Pembrolizumab 200 mg is administered IV once as monotherapy, 14 days after the initiation of High dose cytarabine (HiDAC) salvage induction chemotherapy. Subjects who have a response to induction phase will receive maintenance pembrolizumab at 200 mg IV every 3 weeks for up to 2-years of maintenance therapy (beginning on day 1 of maintenance).Subjects who are ineligible for pembrolizumab administration by day 21 will be removed from the study.
Period: Overall Study
Arm/Group | Single Arm Pembrolizumab
Started | 38
Completed | 37
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: One subject is excluded from the analysis population due to an adverse event from the standard of care high dose cytarabine and did not receive any of the treatment of interest (pembrolizumab).
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 54 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 37
Acute myeloid leukemia (AML) type [Count of Participants; unit: Participants] — Acute myeloid leukemia (AML) is considered to be "refractory" in patients who do not respond to intensive induction chemotherapy. Relapsed AML is the return of leukemia cells after a patient has reached complete remission
  Participants
    Refractory AML | 16
    Relapsed AML | 21
Risk [Count of Participants; unit: Participants] — European LeukemiaNet (ELN) 2017 genetic risk stratification
  Participants
    Favorable | 6
    Intermediate | 12
    Adverse | 19
Secondary Acute Myeloid Leukemia (AML) [Count of Participants; unit: Participants] | 13
Median Bone Marrow Blast Percentage [Median (Full Range); unit: percentage of blast cells] | 28 [6 to 94]

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Complete Remission (CR)
Description: The rate of overall CR includes CR and CR with incomplete recovery (CRi) as defined by the International European LeukemiaNet Guidelines in AML. CR is defined as bone marrow blasts <5%; absence of Auer rods; absence of extramedullary disease; absolute neutrophil count >1,000/microliter (mcL); platelet count >100,000/mcL; independence of red cell transfusions and CRi is defined as meeting all CR criteria except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL) plus independent of platelet transfusions.
Time Frame: Day 14 until 2 years complete on study treatment and after full hematologic recovery from HiDAC followed by pembrolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Participants | 14

2. Secondary Outcome: Rate of Unacceptable Toxicity
Description: number of participants with drug-related grade 3 (severe) non-hematologic toxicity (with exception of infusion reactions, rash, fever, infection, nausea, fatigue, and anorexia) persisting for >7 days with supportive care, or any drug-related non-hematologic grade >4 (life-threatening) toxicity (excluding infection). Toxicity will be classified and graded according to National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term ranging from 1 (mild) to 5 (death related to adverse event).
Time Frame: Day 14 until 2 years complete on study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Participants | 0

3. Secondary Outcome: Objective Overall Response Rate: Partial Remission (PR) + Complete Remission (CR) + Complete Remission With Incomplete Blood Count Recovery (CRi) for HiDAC Followed by Pembrolizumab
Description: PR+CR+CRi as determined by International European LeukemiaNet Guidelines in AML. PR is defined as bone marrow blasts 5-25% and decrease of pretreatment bone marrow blast % by >50%; all hematologic criteria of CR. CR is defined as bone marrow blasts <5%; absence of Auer rods; absence of extramedullary disease; absolute neutrophil count >1,000/microliter (mcL); platelet count >100,000/mcL; independence of red cell transfusions and CRi is defined as meeting all CR criteria except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL) plus independent of platelet transfusions.
Time Frame: Day 14 until 2 years complete on study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Participants | 16

4. Secondary Outcome: Median Relapse-free Survival (RFS) of Patients Receiving Maintenance Pembrolizumab
Description: RFS will be defined as time from day 1 of Complete Remission (CR) or Complete Remission With Incomplete Blood Count Recovery (CRi) to relapse or death from any cause. CR is defined as bone marrow blasts <5%; absence of Auer rods; absence of extramedullary disease; absolute neutrophil count >1,000/microliter (mcL); platelet count >100,000/mcL; independence of red cell transfusions and CRi is defined as meeting all CR criteria except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL) plus independent of platelet transfusions.
Time Frame: from Day 1 of complete remission up to 7 years of follow-up (a median of 7.8 months of survivor follow-up at time of reporting)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Months | 6.9 [4.2 to 11.5]

5. Secondary Outcome: Median Progression-free Survival (PFS) of Patients Receiving Maintenance Pembrolizumab.
Description: PFS will be defined as time from day 1 of response (i.e., PR/CR/CRi) to progression or death from any cause. PR+CR+CRi s determined by International European LeukemiaNet Guidelines in AML. PR is defined as bone marrow blasts 5-25% and decrease of pretreatment bone marrow blast % by >50%; all hematologic criteria of CR. CR is defined as bone marrow blasts <5%; absence of Auer rods; absence of extramedullary disease; absolute neutrophil count >1,000/microliter (mcL); platelet count >100,000/mcL; independence of red cell transfusions and CRi is defined as meeting all CR criteria except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL) plus independent of platelet transfusions.
Time Frame: from Day 1 of response up to 7 years of follow-up (a median of 7.8 months of survivor follow-up at time of reporting)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Months | 5.7 [1.9 to 7.3]

6. Secondary Outcome: Median Overall Survival (OS) of Patients Who Received Induction Phase of Treatment.
Description: OS is defined as time from day 1 of treatment until date of last known follow up or death of any cause
Time Frame: from Day 1 of treatment up to 7 years of follow-up (with a median of 7.8 months of follow-up at time of reporting)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm Pembrolizumab
Number analyzed (Participants) | 37
Months | 8.9 [6.0 to 13.1]

ADVERSE EVENTS:
Time Frame: Day 14 until 2 years complete on study treatment
Arm/Group | Single Arm Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 32/37
Serious Adverse Events (participants affected / at risk) | 14/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Pembrolizumab (N=37)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Arachnoiditis (Nervous system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood and lymphatic system disorders - Other, specify -E.Coli infection in blood (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 2
Catheter related infection (Infections and infestations) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Fever (General disorders) | 1
Hypotension (Vascular disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lung infection (Infections and infestations) | 4
Meningitis (Infections and infestations) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Transient ischemic attacks (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Pembrolizumab (N=37)
Abdominal pain (Gastrointestinal disorders) | 8
Acidosis (Metabolism and nutrition disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 5
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 22
Alkaline phosphatase increased (Investigations) | 21
Alkalosis (Metabolism and nutrition disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 32
Anorexia (Metabolism and nutrition disorders) | 11
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Ascites (Gastrointestinal disorders) | 2
Aspartate aminotransferase increased (Investigations) | 23
Ataxia (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Blood bilirubin increased (Investigations) | 18
Blurred vision (Eye disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 5
Cardiac troponin I increased (Investigations) | 3
Catheter related infection (Infections and infestations) | 3
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 6
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Creatinine increased (Investigations) | 9
Cytokine release syndrome (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 16
Dizziness (Nervous system disorders) | 8
Dry eye (Eye disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysarthria (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2
Edema limbs (General disorders) | 6
Edema trunk (General disorders) | 4
Ejection fraction decreased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 3
Enterocolitis infectious (Infections and infestations) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Esophagitis (Gastrointestinal disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Eye pain (Eye disorders) | 4
Facial pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 24
Fever (General disorders) | 22
Flatulence (Gastrointestinal disorders) | 1
Floaters (Eye disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Genital edema (Reproductive system and breast disorders) | 2
Haptoglobin decreased (Investigations) | 1
Headache (Nervous system disorders) | 21
Heart failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 10
Hemolysis (Blood and lymphatic system disorders) | 1
Hepatic infection (Infections and infestations) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 10
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 5
Hyperthyroidism (Endocrine disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 31
Hypocalcemia (Metabolism and nutrition disorders) | 29
Hypokalemia (Metabolism and nutrition disorders) | 29
Hypomagnesemia (Metabolism and nutrition disorders) | 19
Hyponatremia (Metabolism and nutrition disorders) | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Hypotension (Vascular disorders) | 9
Hypothermia (General disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
INR increased (Investigations) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 4
Infusion related reaction (General disorders) | 5
Insomnia (Psychiatric disorders) | 6
Investigations - Other, specify (Investigations) | 8
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Lipase increased (Investigations) | 1
Lung infection (Infections and infestations) | 10
Lymphocyte count decreased (Investigations) | 30
Lymphocyte count increased (Investigations) | 1
Memory impairment (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Mitral valve disease (Cardiac disorders) | 1
Mucosal infection (Infections and infestations) | 3
Mucositis oral (Gastrointestinal disorders) | 5
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Nausea (Gastrointestinal disorders) | 24
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutrophil count decreased (Investigations) | 29
Non-cardiac chest pain (General disorders) | 3
Nystagmus (Nervous system disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Oral pain (Gastrointestinal disorders) | 7
Pain (General disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Photophobia (Eye disorders) | 2
Platelet count decreased (Investigations) | 34
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Prostatic pain (Reproductive system and breast disorders) | 1
Proteinuria (Renal and urinary disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 16
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18
Rectal pain (Gastrointestinal disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 2
Sinus bradycardia (Cardiac disorders) | 2
Sinus pain (Nervous system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 8
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Small intestinal mucositis (Gastrointestinal disorders) | 1
Somnolence (Nervous system disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Tricuspid valve disease (Cardiac disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2
Typhlitis (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Uterine pain (Reproductive system and breast disorders) | 1
Vaginal infection (Infections and infestations) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Vomiting (Gastrointestinal disorders) | 11
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 2
Weight loss (Investigations) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02768792/Prot_SAP_000.pdf